CLINICAL TRIAL: NCT00668902
Title: Rapid Screening Phenotype Test To Evaluate CYP 2C19 Enzyme Activity Using Stable Isotope [13C]Pantoprazole
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Collaborators: Sponsor Name Pending (Industry)
Responsible Party: Principal Investigator, Zeruesenay Desta, Associate Professor of Medicine, Indiana University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 0611-07
Record Dates: First submitted 2008-01-17; First posted 2008-04-29 (Estimated); Results first posted 2014-12-17 (Estimated); Last update posted 2014-12-17 (Estimated); Status verified 2014-12

CONDITIONS: Healthy
Keywords: CYP2C19; Pantoprazole; Genotype; Pharmacokinetics; Metabolism

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- EM of CYP2C19 (Experimental): CYP2C19 enzyme activity in extensive metabolizers of CYP2C19 (CYP2C19*1/*1 genotype, or wild type) was measured by 13C)Pantoprazole breath test.
  Interventions: Drug: [13C]Pantoprazole
- IM of CYP2C19 (Experimental): CYP2C19 activity in heterozygous for deficient CYP2C19 alleles (*2 and *3, IM of CYP2C19) was measured by (13C)Pantoprazole breath test.
  Interventions: Drug: [13C]Pantoprazole
- PM of CYP2C19 (Experimental): Homozygous for CYP2C19 null alleles (*2/*2, *2/*3 or *3/*3, Poor metabolizers) was measured by (13C)Pantoprazole breath test.
  Interventions: Drug: [13C]Pantoprazole

INTERVENTIONS:
Drug: [13C]Pantoprazole — [13C]Pantoprazole was administered to EM, IM and PM of CYP2C19 and enzyme activity was measured through breath test and compared among the genotypes
  Other Names: Breath test

SUMMARY:
The purpose of this study is to determine the function of an enzyme that breaks down drugs and helps the removal of drugs from your body. This enzyme is called cytochrome P450 2C19 and is located in your liver. Exposure to other medications or variations in genes that you have inherited from your parents, may speed up or slow the function of this enzyme. As a result, some patients may develop unwanted effects from a drug while some other patients may not get benefit from taking the same drug. The aim of this study is to determine the function of this enzyme in your liver. We will do this by performing a series of breath tests and blood samples after you take pantoprazole. Pantoprazole is approved as an oral and intravenous drug by the Food and Drug Administration (FDA).

DETAILED DESCRIPTION:
The goal of this study is to develop a quick and reliable method that will diagnose hepatic CYP2C19 function and could be used routinely in clinical practice. Specifically, we propose to test pantoprazole - 13C as a probe for determining CYP2C19 phenotype. Pantoprazole, 5-(difluoromethoxy)-2-[[(3,4-dimethoxy-2-pyridyl)-methyl]sulfinyl]-1H -benzimidazole, is a substituted benzimidazole sulfoxide and a selective and long-acting proton pump inhibitor. This drug is widely used clinically in the treatment of severe gastroesophageal reflux disease, and for treatment of duodenal and gastric ulceration. Pantoprazole is extensively metabolized in the liver, with almost 80% of an oral or intravenous dose is excreted as metabolites in urine. The main metabolite is formed by O-demethylation at the 4-position of the pyridine ring by CYP2C19, followed by conjugation with sulphate (M2), while pantoprazole sulfone formed by CYP3A represents a minor metabolic pathway(20). The critical role of CYP2C19 in the in vivo clearance of the drugs is further demonstrated by the fact that healthy volunteers that are PMs of this enzyme achieve approximately 6-fold higher pantoprazole exposure than those who are extensive metabolizers of CYP2C19(20). This concept proposal exploits the use of the 13C-label that is incorporated at the O-methyl site of pantoprazole, which specifically designed for the CYP2C19-mediated O-demethylation (Figure 1). Then, during catalysis, CYP2C19-pantoprazole reaction in the liver results in the release of 13CO2 which is then eliminated from the body via the lung expired breath. The subsequent quantification of 13CO2 allows indirect determination of the hepatic CYP2C19 enzyme and thus the pharmacokinetics of its substrates. The salient features of the 13C-breath test means that this test would be non-invasive, non-radioactive, safe and simple. The protocol in general can be performed rapidly (one hour or less after pantoprazole administration) and can be determined directly at the point of care (e.g., hospitals and physicians' offices) using relatively inexpensive instrumentation (UBiT-IR300IR spectrometer; Meretek), and patients do not require waiting for hours or days for diagnostic results. This test may be particularly important to probe the activity of CYP2C19 for infants, children, pregnant and lactating women, seniors averse to the use of needles or in poor health and subjects scared of blood draws.

ELIGIBILITY:
Inclusion Criteria:

1. Asian male or female subjects between 18 and 49 years of age, who are in good physical health with no significant medical problems or laboratory test abnormalities. Subjects should have normal liver and kidney function.
2. Subjects with BMI <30 which will be determined by Metropolitan height and weight tables. Subjects must weigh at least 110 pounds.
3. Subjects must agree to refrain from taking any prescription and over-the-counter medications, as well as any herbal medications one week before the start of the study and during the study period.
4. Subjects must agree to refrain from consuming alcohol 48 hours before the start of the study and during the study period.
5. Subjects must be capable of satisfying protocol requirements and be able to sign written informed consent.

Exclusion Criteria:

1. Subjects who have a history of intolerance or allergy to the study drug: pantoprazole.
2. Subjects who have donated blood within the last 60 days of the screening visit or plan to donate blood during the course of the study or within 60 days after study completion.
3. Subjects who have had treatment with any investigational drug within the past 30 days.
4. Subjects who have used illegal drugs within three months prior to enrollment.
5. Female subjects currently taking oral contraceptive birth control pills and who are unwilling or unable to stop oral contraceptives and use a barrier contraceptive method (such as condom, contraceptive foams, etc.) starting from the time of screening phase to the completion of the study.
6. Female subjects who are pregnant or lactating.
7. Subjects who are unreliable in the opinion of the study physician.

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2007-03; Primary Completion 2008-12 (Actual); Study Completion 2009-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Zeruesenay Desta, PhD, Principal Investigator — Indiana University
Locations (1):
- Indiana University, Indianapolis, Indiana, United States

REFERENCES:
- [Background] Desta Z, Zhao X, Shin JG, Flockhart DA. Clinical significance of the cytochrome P450 2C19 genetic polymorphism. Clin Pharmacokinet. 2002;41(12):913-58. doi: 10.2165/00003088-200241120-00002. PMID 12222994
- [Background] Goldstein JA. Clinical relevance of genetic polymorphisms in the human CYP2C subfamily. Br J Clin Pharmacol. 2001 Oct;52(4):349-55. doi: 10.1046/j.0306-5251.2001.01499.x. PMID 11678778
- [Background] De Morais SM, Wilkinson GR, Blaisdell J, Meyer UA, Nakamura K, Goldstein JA. Identification of a new genetic defect responsible for the polymorphism of (S)-mephenytoin metabolism in Japanese. Mol Pharmacol. 1994 Oct;46(4):594-8. PMID 7969038
- [Background] de Morais SM, Wilkinson GR, Blaisdell J, Nakamura K, Meyer UA, Goldstein JA. The major genetic defect responsible for the polymorphism of S-mephenytoin metabolism in humans. J Biol Chem. 1994 Jun 3;269(22):15419-22. PMID 8195181
- [Background] Ibeanu GC, Blaisdell J, Ghanayem BI, Beyeler C, Benhamou S, Bouchardy C, Wilkinson GR, Dayer P, Daly AK, Goldstein JA. An additional defective allele, CYP2C19*5, contributes to the S-mephenytoin poor metabolizer phenotype in Caucasians. Pharmacogenetics. 1998 Apr;8(2):129-35. doi: 10.1097/00008571-199804000-00006. PMID 10022751
- [Background] Ibeanu GC, Goldstein JA, Meyer U, Benhamou S, Bouchardy C, Dayer P, Ghanayem BI, Blaisdell J. Identification of new human CYP2C19 alleles (CYP2C19*6 and CYP2C19*2B) in a Caucasian poor metabolizer of mephenytoin. J Pharmacol Exp Ther. 1998 Sep;286(3):1490-5. PMID 9732415
- [Background] Ferguson RJ, De Morais SM, Benhamou S, Bouchardy C, Blaisdell J, Ibeanu G, Wilkinson GR, Sarich TC, Wright JM, Dayer P, Goldstein JA. A new genetic defect in human CYP2C19: mutation of the initiation codon is responsible for poor metabolism of S-mephenytoin. J Pharmacol Exp Ther. 1998 Jan;284(1):356-61. PMID 9435198
- [Background] Sim SC, Risinger C, Dahl ML, Aklillu E, Christensen M, Bertilsson L, Ingelman-Sundberg M. A common novel CYP2C19 gene variant causes ultrarapid drug metabolism relevant for the drug response to proton pump inhibitors and antidepressants. Clin Pharmacol Ther. 2006 Jan;79(1):103-13. doi: 10.1016/j.clpt.2005.10.002. PMID 16413245

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | EM of CYP2C19 | IM of CYP2C19 | PM of CYP2C19
Started | 10 | 10 | 5
Completed | 10 | 10 | 5
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | EM of CYP2C19 | IM of CYP2C19 | PM of CYP2C19 | Total
Number analyzed (Participants) | 10 | 10 | 5 | 25
Age, Continuous [Mean (Standard Deviation); unit: years] | 26.2 (5.3) | 26.4 (6.1) | 24.3 (3.3) | 25.63 (1.159)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 7 | 2 | 15
  Male | 4 | 3 | 3 | 10
Region of Enrollment [Number; unit: participants]
  United States | 10 | 10 | 5 | 25
BMI [Mean (Standard Deviation); unit: kg/m^2] | 24.8 (3.6) | 24.8 (3.5) | 23 (1.3) | 24.2 (1.039)

OUTCOME MEASURES:

1. Primary Outcome: DOBmax (Maximum Value of DOB)
Description: The stable isotope [13C]pantoprazole is O-demethylated by cytochrome P450 CYP2C19 and that the 13CO2 produced and exhaled in breath as a result can serve as a safe, rapid, and noninvasive phenotyping marker of CYP2C19 activity in vivo.
  Exhaled 13CO2 and 12CO2 were measured by IR spectroscopy before (baseline) and 2.5 to 120 min after dosing. Ratios of 13CO2/12CO2 after [13C]pantoprazole relative to 13CO2/12CO2 at baseline were expressed as change over baseline (DOB).
Time Frame: baseline and 2.5, 5, 10, 15, 20, 25, 30, 40, 50, 60, 90, and 120 min after dosing
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | EM of CYP2C19 | IM of CYP2C19 | PM of CYP2C19
Number analyzed (Participants) | 10 | 10 | 5
ratio | 4.44 (1.79) | 3.49 (1.18) | 0.92 (0.18)

ADVERSE EVENTS:
Arm/Group | EM of CYP2C19 | IM of CYP2C19 | PM of CYP2C19
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10 | 0/5
Other Adverse Events (participants affected / at risk) | 0/10 | 0/10 | 0/5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No